CLINICAL TRIAL: NCT00427297
Title: Optimizing Pediatric HIV-1 Treatment in Infants With Prophylactic Exposure to Nevirapine, Nairobi, Kenya (6-12 Month RCT)
Brief Title: Optimizing Pediatric HIV-1 Treatment in Infants With Prophylactic Exposure to Nevirapine, Nairobi, Kenya
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: There is no longer equipoise. DSMB recommended termination.
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, Global Health, Medicine, Epidemiology, Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002049; 2R01HD023412-16 (NIH); 06-1886-D 02
Record Dates: First submitted 2007-01-22; First posted 2007-01-29 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Pediatric; nevirapine; HAART; Resistance; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Stavudine; abacavir, lamivudine drug combination; Didanosine; abacavir; Nevirapine; efavirenz; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NVP-containing (Experimental): Infants randomized to this arm will receive nevirapine-containing HAART regimen
  Interventions: Drug: AZT/3TC/NVP (zidovudine/lamivudine/nevirapine); Drug: d4T/3TC/NVP (stavudine/lamivudine/nevirapine); Drug: ABC/3TC/NVP (abacavir/lamivudine/nevirapine)
- NVP-sparing (Active Comparator): Infants randomized to this arm will receive nevirapine-sparing HAART
  Interventions: Drug: AZT/3TC/ABC (zidovudine/lamivudine/abacavir); Drug: d4T/3TC/ABC (stavudine/lamivudine/abacavir); Drug: ddI/ABC/LPV/r (didanosine/abacavir/lopinavir-ritonavir); Drug: ABC/ ddI or TDF / NVP or EFV (abacavir / didanosine or tenofovir / nevirapine or efavirenz)

INTERVENTIONS:
Drug: AZT/3TC/NVP (zidovudine/lamivudine/nevirapine) — First line regimen
  Arms: NVP-containing
Drug: d4T/3TC/NVP (stavudine/lamivudine/nevirapine) — First line regimen
  Arms: NVP-containing
Drug: AZT/3TC/ABC (zidovudine/lamivudine/abacavir) — First line regimen
  Arms: NVP-sparing
Drug: d4T/3TC/ABC (stavudine/lamivudine/abacavir) — First line regimen For children who have anaemia(Hb of<8g/dl), AZT will be substituted for d4T.
  Arms: NVP-sparing
Drug: ddI/ABC/LPV/r (didanosine/abacavir/lopinavir-ritonavir) — Second line regimen
  Arms: NVP-sparing
Drug: ABC/ ddI or TDF / NVP or EFV (abacavir / didanosine or tenofovir / nevirapine or efavirenz) — Second line regimen - Among children randomized to NVP sparing HAART, who will be initiated on a regimen containing lopinavir/ritonavir, zidovudine and lamivudine will be substituted with abacavir and didanosine or tenofovir (TDF) and lopinavir/ ritonavir will be replaced with nevirapine or efavirenz (EFV) in case of treatment failure of the LPV/r containing regimen.
  Arms: NVP-sparing
Drug: ABC/3TC/NVP (abacavir/lamivudine/nevirapine) — First line regimen
  Arms: NVP-containing

SUMMARY:
Globally, children who acquire HIV-1 increasingly do so in the context of maternal antiretroviral prophylaxis. It is important to determine whether maternal antiretroviral prophylaxis should alter infant treatment regimens. Nevirapine (NVP) is commonly used for PMTCT and is also a commonly used first-line drug for treatment of pediatric HIV-1. Approximately half of infants exposed to NVP have detectable NVP resistance early in infancy, with loss of detectable resistance over time. Thus, if an HIV-1 infected child was exposed to single-dose NVP prophylaxis, the question remains whether NVP or any NNRTI can be used effectively in therapeutic regimens. Alternative PI-based regimens are associated with heat-lability, poor palatability, cumulative toxicity, and fewer salvage options. This poses challenges for pediatric PI-based highly active antiretroviral therapy (HAART) in settings without refrigeration and limited antiretroviral repertoire. It is plausible that in older NVP-exposed infants (older than 6 months since exposure) who are genotypically NVP-susceptible, that nevirapine will be effective and useful.

We propose to study resistance in a pediatric HIV-1 clinical trial involving 100 children. Among children enrolled at between 6 and 18 months of age, we will provide real-time field-based genotypic NVP-resistance testing, and randomize 100 NVP-susceptible children to NVP-containing versus NVP-sparing HAART to compare therapeutic response, adverse events, and morbidity in the 2 arms during 2-year follow-up. Follow-up in these studies will be closely monitored by an external Data Safety and Monitoring Board (DSMB).

DETAILED DESCRIPTION:
Hypotheses

1. Infants older than 6 months who do not have detectable nevirapine resistance on genotypic testing will respond equivalently to a nevirapine-sparing or a nevirapine-containing HAART regimen, despite previous single-dose nevirapine exposure.
2. Genotypic drug resistance levels may predict response to therapy and clinical progression.

Specific Aims/Primary Objectives

1. To compare response to therapy (viral levels, CD4%, growth, and morbidity) in infants without detectable nevirapine-resistance on population-based sequencing who are randomized to nevirapine-containing versus nevirapine-sparing HAART.
2. To develop methods to detect and quantify nevirapine resistance mutations present at low frequency in the virus population in order to examine the relationship between the copy number of such variants and virologic failure of infants treated with nevirapine-containing HAART.

Secondary Aim/Secondary Objective: To determine predictors of non-progression in these studies, including: age, time since nevirapine-exposure, adherence, HIV-1 specific immune responses, baseline HIV-1 RNA, CD4 percent, and immune activation.

Design: Randomized clinical trial in which infant 6-18 months of age will be randomized to nevirapine containing versus nevirapine sparing HAART regimen and followed for 24 months.

Population: HIV-1 infected infants (6-12 months) meeting eligibility will be enrolled. Infants who were exposed to nevirapine in-utero or following delivery, with no detectable resistance to nevirapine will be eligible for enrollment.

Sample size: 100 infants will be enrolled (50 infants in each arm).

Treatment: All infants will be treated with NVP containing or sparing HAART. The regimen will be prescribed according to WHO and Kenyan national guidelines on dosage and combination of antiretroviral drugs. The HAART regimen that will be used in this study are:

First line regimen:

For infants on NVP containing HAART

* AZT/3TC/NVP (zidovudine/lamivudine/nevirapine)
* d4T/3TC/NVP (stavudine/lamivudine/nevirapine)
* ABC/3TC/NVP (abacavir/lamivudine/nevirapine)

For infants on NVP sparing HAART

* AZT/3TC/ABC (zidovudine/lamivudine/abacavir)
* d4T/3TC/ABC (stavudine/lamivudine/abacavir)

For children who have anaemia (Hb of <8g/dl), AZT will be substituted for d4T.

Second line regimen:

* ddI/ABC/LPV/r (didanosine/abacavir/lopinavir-ritonavir (kaletra))
* ABC / ddI or TDF / NVP or EFV (abacavir / didanosine or tenofovir / nevirapine or efavirenz) Among children randomized to NVP sparing HAART, who will be initiated on a regimen containing lopinavir/ritonavir, zidovudine and lamivudine will be substituted with abacavir and didanosine or tenofovir (TDF) and lopinavir/ ritonavir will be replaced with nevirapine or efavirenz (EFV) in case of treatment failure of the LPV/r containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 months age
* HIV-1 DNA detection with confirmation (positive on two HIV-1 DNA filter paper tests)
* Mother exposed to NVP-containing PMTCT regimen during currently ended pregnancy and/or infant received NVP-containing PMTCT regimen
* Infant susceptible to NVP (i.e. no detectable NVP resistance on genotypic testing)
* Caregiver of infant plans to reside in Nairobi for at least 3 years
* Caregiver is able to provide sufficient location information

Exclusion Criteria:

* Infant has received any prior antiretroviral therapy (expect prophylaxis for PMTCT)
* Infant has evidence of active tuberculosis
* Mother currently receiving NVP-containing HAART and breastfeeding the infant

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace C John-Stewart, MD, PhD, Principal Investigator — University of Washington; Dalton Wamalwa, MMed, MPH, Principal Investigator — Department of Paediatrics and Child Health, Kenyatta National Hospital, University of Nairobi
Locations (1):
- Kenyatta National Hospital, University of Nairobi, Nairobi, Kenya

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NVP-containing | NVP-sparing
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVP-containing | NVP-sparing | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 7 [6 to 10] | 8 [6 to 10] | 7 [6 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 9 | 10 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 17 | 17 | 34
CD4% [Median (Inter-Quartile Range); unit: percentage of cells] | 22 [14 to 29] | 18 [13 to 25] | 21.5 [13 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Mortality
Description: Death during follow-up
Time Frame: 2 years
Population: Analysis was conducted at DSMB termination of study with 15.6 person-years of follow-up time in the cohort overall; 8.5 person-years in NVP-containing and 7.1 person-years in NVP-sparing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | NVP-containing | NVP-sparing
Number analyzed (Participants) | 17 | 17
Participants | 4 | 5

2. Primary Outcome: Immunologic Failure
Description: Immunologic treatment failure was defined as CD4% dropping below 15%, after a previous result greater than or equal to 15% (following along WHO Guidelines).
Time Frame: 2 years
Population: 15.6 person years of follow-up overall at time of DSMB closure of study
Measure: Count of Participants; unit: Participants
Arm/Group | NVP-containing | NVP-sparing
Number analyzed (Participants) | 12 | 13
Participants | 2 | 1

3. Primary Outcome: Viral Failure
Description: Virologic treatment failure was defined as follow-up (at least 24 weeks after enrollment date) viral load > 400 copies.
Time Frame: 2 years
Population: 15.6 person years of follow-up overall at time of DSMB closure of study
Measure: Count of Participants; unit: Participants
Arm/Group | NVP-containing | NVP-sparing
Number analyzed (Participants) | 8 | 5
Participants | 2 | 2

4. Secondary Outcome: Incidence of Severe Adverse Events (Excluding Mortality)
Time Frame: 2 years
Population: 15.6 person-years of follow-up overall at time of DSMB closure of study
Measure: Number; unit: event
Arm/Group | NVP-containing | NVP-sparing
Number analyzed (Participants) | 17 | 17
event | 21 | 6

ADVERSE EVENTS:
Time Frame: 2 years
Description: 15.6 person years overall of follow-up at time of DSMB closure of study
Groups:
- NVP-containing: NVP-containing (AZT/3TC/NVP; d4T/3TC/NVP; or ABC/3TC/NVP) antiretroviral triple combination therapy.
  Second-line regimens based on the WHO pediatric treatment guidelines, 2006.
- NVP-sparing: NVP-sparing (AZT/3TC/LPV/r; or d4T/3TC/LPV/r1) antiretroviral triple combination therapy.
  Second-line regimens based on the WHO pediatric treatment guidelines, 2006.
Arm/Group | NVP-containing | NVP-sparing
All-Cause Mortality (participants affected / at risk) | 4/17 | 5/17
Serious Adverse Events (participants affected / at risk) | 4/17 | 3/17
Other Adverse Events (participants affected / at risk) | 13/17 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVP-containing (N=17) | NVP-sparing (N=17)
Pneumonia or respiratory (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hepatotoxicity (Hepatobiliary disorders) | 2 | 1
Severe anemia (Blood and lymphatic system disorders) | 2 | 0
Hyperamylasemia (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVP-containing (N=17) | NVP-sparing (N=17)
Rash (Skin and subcutaneous tissue disorders) | 3 | 7
Gastroenteritis (Gastrointestinal disorders) | 4 | 4
Milestone regression (Nervous system disorders) | 1 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 | 5

LIMITATIONS AND CAVEATS:
The study team suggested discontinuation of the trial and the DSMB concurred based on slow accrual and based on new data that emerged after the RCT was initiated which made the trial question less relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No